CLINICAL TRIAL: NCT05837039
Title: A Comparison of Healthcare Provider and Caregiver Perception of Discomfort in Advanced Cancer Patients Who Have a Hypoactive Delirium
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-1177; NCI-2022-02412 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-04-17; First posted 2023-05-01 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Hypoactive Delirium
MeSH Terms: interventions — Health Personnel

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare Provider and Caregiver Perception of Discomfort: Participants will be providing demographic information about you (age, sex/gender, race, ethnicity, educational level, if the participant are in the same household as the patient, if participants are the primary caregiver of the patient, and whether you live in a rural, suburban, or urban environment) Your feelings about your loved one's comfort level Your feelings about symptoms you think affect comfort level Behaviors seen while at the bedside of your loved one
  Interventions: Behavioral: Healthcare Provider; Behavioral: Caregiver Perception

INTERVENTIONS:
Behavioral: Healthcare Provider — Questionnaires
Behavioral: Caregiver Perception — Questionnaires

SUMMARY:
To learn about your feelings as a caregiver about the level of discomfort of patients who have hypoactive delirium (loss of contact and response to reality) and who are at the end of life

DETAILED DESCRIPTION:
Primary Objective:

To assess the caregiver's perception of the level of discomfort of patients who have a hypoactive delirium and who are considered actively dying. The caregiver's perception will be based upon the Caregiver Survey of Patient Discomfort.

Secondary Objective:

To compare the perception of discomfort between the caregiver and bedside nurse. The caregiver's perception will be based upon the Caregiver Survey of Patient Discomfort, and the nurse's perception will be based upon the Healthcare Provider Survey of Patient Discomfort.

Exploratory Objective:

To assess associations between patient demographics and clinical characteristics as well as caregiver and nurse demographics on corresponding caregiver and nurse survey responses.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Patients with advanced cancer. Advanced cancer is defined as locally invasive, metastatic or recurrent cancer. Hematologic malignancies will also be included.
2. Patients who are admitted to the acute palliative care unit (APCU) at MD Anderson Cancer Center.
3. Patients who are unable to respond to questioning in the past 24 hours as determined by the attending physician, fellow physicians, or nursing staff of the APCU.
4. Patients who are considered to be actively dying, as defined as likely to die during the admission and not regain consciousness. The physical exam findings that will be utilized to help define those patients who are actively dying may include one but not limited to one of the following symptoms: pulseless of the radial artery, Cheyne-stokes breathing, peripheral cyanosis, apnea periods, respiration with mandibular movement, turbulent airway noise produced on inspiration and/or expiration due to airway secretions commonly known as the "death rattle", and loss of nasolabial folds The presence of these signs will be based on the reporting of the attending physician, fellow physicians or nursing staff of the APCU.
5. Patients who have an unpaid adult caregiver at bedside age 18 years or older, who is willing and able to provide informed consent and who has been present at bedside for at least 3 hours a day.

Patient Exclusion Criteria:

1. Patients who had a hyperactive or mixed delirium in which they either had high level of arousal due to delirium or had mixed episodes of arousal and agitation with periods of unresponsiveness.
2. A family member or caregiver who cannot provide informed consent, or who cannot speak and read English.

Caregiver Inclusion Criteria:

1. Unpaid adult caregiver at bedside age 18 years or older, who is willing and able to provide informed consent, able to speak and read English, and who has been present at bedside for at least 3 hours a day.

Nursing Provider Inclusion Criteria:

1. Nursing providers in the acute palliative care unit who are providing direct patient care to eligible patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: M D Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Likert Scale Survey | through study completion; an average of 1 year.
  Score Scales: (1-5)
  1. Strongly Disagree
  2. Disagree
  3. Neither Agree Nor Disagree
  4. Agree
  5. Strongly Agree

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tang, MD, Principal Investigator — University of M D Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org